CLINICAL TRIAL: NCT02041923
Title: Feeding and Transition to Home for Preterms at Social Risk
Acronym: H-HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rosemary White-Traut, Professor (retired), University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-0139; 1R01HD050738 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Premature Birth
Keywords: preterm infant; stable infant; mother-infant interaction; health care cost; H-HOPE intervention; mother outcomes; infant behavioral organization; infant growth
MeSH Terms: conditions — Premature Birth | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Control (Placebo Comparator): Mothers received equal amount of attention from the team. Attention consisted of additional teaching regarding premature infant care.
  Interventions: Other: Attention Control
- H-HOPE Intervention (Experimental): H-HOPE was administered twice daily by the mother.
  Interventions: Behavioral: H-HOPE

INTERVENTIONS:
Behavioral: H-HOPE — Infant remediation using a developmentally appropriate multisensory intervention addresses the specific behavioral organization needs of premature infants. Maternal redefinition and re-education by a nurse-community advocate team uses participatory guidance to address the needs of mothers of premature infants.
  Other Names: ATVV Intervention
  Arms: H-HOPE Intervention
Other: Attention Control — Mothers received equal amount of attention from the team. Attention consisted of additional teaching regarding premature infant care.
  Other Names: Education
  Arms: Attention Control

SUMMARY:
Premature infants are at high risk of suboptimal health and development. This randomized clinical trial evaluated the impact of a developmentally based intervention, H-HOPE (Hospital-home transition: optimizing prematures' environment), for infants born between 29-34 weeks gestational age (GA) with at least two social-environmental risk factors. H-HOPE will improve infant behavior, mother care for the infants, mother-infant interaction and will reduce health care costs.

DETAILED DESCRIPTION:
Premature infants are at high risk of suboptimal health and development. This randomized clinical trial evaluated the impact of a developmentally based intervention, H-HOPE (Hospital-home transition: optimizing prematures' environment), for infants born between 29-34 weeks gestational age (GA) with at least two social-environmental risk factors. H-HOPE is innovative because it integrates two components used successfully in prior research but never before combined. Infant remediation using a developmentally appropriate multisensory intervention addresses the specific behavioral organization needs of premature infants. Maternal redefinition and re-education by a nurse-community advocate team uses participatory guidance to address the needs of mothers of premature infants. The synergistic effect of these simultaneous improvements for infant and mother should lead to: 1) more mature infant behavioral organization and hospital progression; 2) improved maternal recognition of infant behavioral cues, greater confidence in infant care, more positive perception of the infant, and lower anxiety; 3) more positive mother-infant interaction and greater mother-infant contingency; 4) improved infant development and growth; and 5) lower infant health care utilization and costs. H-HOPE provides intervention from 32 weeks GA to one month corrected age, a time of transition to oral feeding, from the hospital to home, and from hospital to outpatient providers, when mothers of premature infants express need for support. We will randomly assign 252 infants to the H-HOPE or the Attention Control group. Power analysis shows that with an 80% retention rate, we will have adequate power to identify expected intervention effects. Variables are measured during hospital stay, at intake, immediately prior to discharge, and at six weeks corrected age. Analyses employ Hierarchical Linear Modeling clustered within clinical sites, with infant sex, biologic and social-environmental risk factors as covariates. If successful, H-HOPE will provide a national model for improving early infant health and development and reducing health costs. For example, reducing hospital stays by just three days for the almost 500,000 infants born prematurely could save over two billion dollars annually.

ELIGIBILITY:
Inclusion Criteria:

29-34 weeks gestation at birth

no other major health problems

mothers have at least 2 socio-environmental risk factors such as African American or Latina

Less then high school education

history of mental illness

less than 150% poverty level

2 children less than 24 months old

4 or more children living in the home

living in a disadvantaged neighborhood

Exclusion Criteria:

Infant has congenital anomaly

Necrotizing enterocolitis

Brain injury

chronic lung disease

prenatal drug exposure

mother is an illicit drug user

mother is not the legal guardian

-

Ages: 2 Hours to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary C. White-Traut, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Mount Sinai Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vonderheid SC, Park CG, Rankin K, Norr KF, White-Traut R. Impact of an integrated mother-preterm infant intervention on birth hospitalization charges. J Perinatol. 2020 Jun;40(6):858-866. doi: 10.1038/s41372-019-0567-7. Epub 2020 Jan 8. PMID 31913324
- [Derived] Arianas EA, Rankin KM, Norr KF, White-Traut RC. Maternal weight status and responsiveness to preterm infant behavioral cues during feeding. BMC Pregnancy Childbirth. 2017 Apr 11;17(1):113. doi: 10.1186/s12884-017-1298-4. PMID 28399825
- See also: Mybiblio — https://www.ncbi.nlm.nih.gov/myncbi/1zuy2pmUXmu5a/bibliography/public/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants and their mothers were screened by the research team. Mothers of eligible infants were approached for consent. We had IRB approval to recruit 230 mother-infants dyads. We recruited 198 total mother-infant dyads.
Pre-assignment Details: Random assignment was conducted after enrollment.
Groups:
- Attention Control: Mothers received equal amount of attention from the team
  H-HOPE: Infant remediation using a developmentally appropriate multisensory intervention addresses the specific behavioral organization needs of premature infants. Maternal redefinition and re-education by a nurse-community advocate team uses participatory guidance to address the needs of mothers of premature infants.
Period: Overall Study
Arm/Group | Attention Control | H-HOPE Intervention
Started | 102 | 96
Completed | 76 | 66
Not Completed | 26 | 30
Not completed — Lost to Follow-up | 26 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | H-HOPE Intervention | Total
Number analyzed (Participants) | 102 | 96 | 198
Age, Continuous [Mean (Standard Deviation); unit: weeks of gestation] | 32 (1.6) | 32 (1.7) | 32 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 59 | 54 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 43 | 90
  Not Hispanic or Latino | 55 | 53 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 55 | 53 | 108
  Race: White | 47 | 43 | 90
  Race: More than one race | 0 | 0 | 0
  Race: Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 55 | 53 | 108
  latino | 47 | 43 | 90
Region of Enrollment [Number; unit: participants]
  United States | 102 | 96 | 198

OUTCOME MEASURES:

1. Primary Outcome: Infant Behavioral Organization
Description: Orally directed behavioral cues (hand to mouth, hand swipes at mouth, sucking on hand, sucking on tongue, tonguing) per week.
Time Frame: From birth to 36 weeks
Measure: Mean (Standard Deviation); unit: Orally directed behavioral cues per week
Groups:
- Attention Control: Mothers received equal amount of attention from the team.
Arm/Group | Attention Control | H-HOPE Intervention
Number analyzed (Participants) | 102 | 96
Orally directed behavioral cues per week | 33.2 (42.4) | 51.8 (56.7)

2. Primary Outcome: Mother-Infant Interaction
Description: Mother-infant interaction during feeding measured via the Nursing Child Assessment Feeding Scale (NCAFS). The NCAFS possible scores ranged from 0-76. A higher score indicates a better outcome.
Time Frame: 34 - 44 weeks postmenstrual age
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Control | H-HOPE Intervention
Number analyzed (Participants) | 76 | 66
units on a scale | 62.5 (7.0) | 64.3 (5.2)

3. Secondary Outcome: Infant Growth
Description: Infant growth in weight gain was measured at entry I into the study and at hospital discharge.
Time Frame: from birth to hospital discharge, up to 9 weeks
Measure: Mean (Standard Deviation); unit: weight in grams
Arm/Group | Attention Control | H-HOPE Intervention
Number analyzed (Participants) | 37 | 36
weight in grams | 2038 (228) | 2051 (284)
Statistical Analysis 1: Comparison: Attention Control vs H-HOPE Intervention; Test type: Equivalence — A t-test was conducted to evaluate equivalency; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 46.3

4. Secondary Outcome: Health Care Utilization
Description: Illness visits within 6 weeks post discharge
Time Frame: Illness visits within 6 weeks post hospital discharge
Population: Infant outpatient illness appointments
Measure: Mean (Standard Deviation); unit: Illness visits
Arm/Group | Attention Control | H-HOPE Intervention
Number analyzed (Participants) | 69 | 78
Illness visits | 15 (2.8) | 10 (1.2)

ADVERSE EVENTS:
Time Frame: No adverse events occurred during participant enrollment and participation - over a 4 month period..
Arm/Group | Attention Control | H-HOPE Intervention
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/96
Other Adverse Events (participants affected / at risk) | 0/102 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No